CLINICAL TRIAL: NCT07346482
Title: Determining the Effect of Midwife-Led Safe Infant Care Training for Pregnant Women on Awareness of Sudden Infant Death Syndrome and Home Accidents
Acronym: Infant Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ayseren Cevik, Principal Investigator,, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 96/160 (14.11.2025)
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Infant Death; Infant Care; Midwifery; Education; Accident at Home
Keywords: infant; infant death; midwifery care; accident; education
MeSH Terms: conditions — Infant Death | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Following the pre-test, the intervention group will receive training on safe infant care. A final test will be administered via telephone in the second week postpartum.
  Interventions: Other: Education
- Control (No Intervention): Standard care (Turkish Ministry of Health Prenatal Care Guide) will be applied during the follow-up care after the pre-test. A final test will be administered via telephone in the second week postpartum.

INTERVENTIONS:
Other: Education — The educational content consists of general information about sudden infant death syndrome and home accidents in children aged 0-3, as well as prevention methods.
  Arms: Experimental

SUMMARY:
This project is a pioneering study in determining the impact of midwife-led safe infant care training for pregnant women on awareness of sudden infant death syndrome (SIDS) and home accidents. Raising awareness and improving women's knowledge about SIDS and home accidents is expected to help reduce preventable infant deaths. If the effectiveness of this training is proven, integrating it into prenatal care programs would be a significant step towards improving maternal and child health.

DETAILED DESCRIPTION:
This research is designed as a randomized controlled experimental study. The research will be conducted in the NST unit located in the Marsa Obstetrics and Gynecology Annex Building of Seyhan State Hospital between the specified dates. It has been determined that 60 participants should be included in the intervention group and 60 in the control group. Primiparous pregnant women ≥32 weeks of gestation will be included in the study. The study will be conducted in two interviews. The pre-test will be administered at the first meeting with the pregnant woman, and the post-test will be administered in the second week postpartum. The independent variables of the study are safe infant care education, and the demographic and obstetric characteristics of the pregnant women. The dependent variables are awareness of sudden infant death syndrome and scores on the home accident awareness scale for mothers. After normality tests are performed, univariate and multivariate analyses appropriate to the data set will be performed, and a significance level of p<0.05 will be considered. The Statistical Programme for Social Science 22 (SPSS) will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being able to speak and understand Turkish
* Being literate
* Being a primiparous pregnant woman (due to the greater need for information) ≥36th week of pregnancy (because it is close to delivery and there is sufficient time to translate what they have learned into behavior)

Exclusion Criteria:

* Diagnosed high-risk pregnancy
* Diagnosed mental health condition
* Having previously received training/course in safe infant care

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 120 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Home Accident Awareness Scale for Mothers | pre-intervention, immediately after the intervention, after 2 week
  Items are scored on a scale of 1-5. As the scale score increases, mothers' awareness of household accidents will increase.
Sudden Infant Death Syndrome Awareness Scale - Mother Form | pre-intervention, immediately after the intervention, after 2 week
  Items are scored on a scale of 1 to 5. As the score obtained from the scale increases, the awareness score decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University Faculty of Health Sciences Department of Midwifery, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No